CLINICAL TRIAL: NCT00066131
Title: Effects of Periodontal Therapy on Preterm Birth
Brief Title: Obstetrics and Periodontal Therapy (OPT) Study
Acronym: OPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0104M94001; NIDCR-DE014338 (Other: NIDCR)
Record Dates: First submitted 2003-08-04; First posted 2003-08-05 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Periodontitis; Infant, Premature
MeSH Terms: conditions — Periodontitis; Premature Birth | interventions — Root Planing; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scaling and root planing (Active Comparator): Scaling and root planing delivered prior to 21 weeks of gestation.
  Interventions: Procedure: Periodontal scaling and root planing; Procedure: Scaling and root planing
- Placebo (No Intervention): Delayed treatment group. Controls monitored clinically from baseline to 29-32 weeks of gestation. Scaling and root planing provided after delivery.

INTERVENTIONS:
Procedure: Periodontal scaling and root planing — Hard and soft tisse deposits (plaque and calculus) are removed from the tooth and tooth root using hand and ultrasonic instruments.
  Other Names: Deep cleaning
  Arms: Scaling and root planing
Procedure: Scaling and root planing — Delivered using hand and powered scalers and with topical or local (injected) anesthetics as needed. Procedures performed over 1 to 4 90-minute visits.
  Arms: Scaling and root planing

SUMMARY:
The purpose of this study is to determine if non-surgical periodontal (gum) treatment can reduce the incidence of preterm birth and low birth weight babies in mothers with periodontitis (gum disease).

DETAILED DESCRIPTION:
Eight hundred sixteen women who are between 13 and 16 weeks pregnant will be enrolled in this trial. Volunteers will be recruited from Hennepin County Medical Center (MN), the Jackson Medical Mall (MS), the University of Kentucky, and Harlem (NY) Hospital. The incidence of preterm birth is higher at these sites than the national average. Subjects will be randomly assigned to receive non-surgical mechanical periodontal therapy (scaling and root planing) either prior to 20 weeks of their pregnancy or soon after delivery. All subjects will be monitored for progressive periodontitis and will be treated immediately regardless of their group assignment. All women will also receive essential dental care to restore caries and treat abscessed teeth. The primary birth outcome is gestational age at birth and the secondary outcome is birthweight. Maternal risk factors for preterm birth and/or intrauterine growth restriction will be used as covariates in the data analysis. The study will also document the effect of periodontal therapy on immune response, systemic markers of inflammation, periodontal infection and clinical periodontal measure.

ELIGIBILITY:
Inclusion

* Be pregnant in the first 13-16 weeks of gestation as determined by menstrual history and obstetrical ultrasound
* Be at least 16 years of age
* Have at least 20 natural teeth,
* Have bleeding on probing (BOP) on at least 35% of all tooth sites
* Have 4 or more teeth with pockets greater than or equal to 4 mm and attachment loss greater than or equal to 2 mm

Exclusion

* Are unable to provide informed consent or are unable to cooperate with the study protocol.
* May be placed at medical risk as a result of participation (i.e. subjects with hematologic disease or other disorders tha preclude routine non-surgical periodontal therapy).
* Have multiple fetuses as diagnosed by ultrasound.
* Require antibiotic prophylaxis for periodontal procedures
* Require greater than 3 essential dental care visits because of extensive decay and/or broken teeth and are likely to have less than 20 natural teeth following essential dental care

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2003-03; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Gestational age at birth | At delivery

SECONDARY OUTCOMES:
Infant birth weight | At delivery
Periodontal probing depth | 29-32 weeks of gestation
Clinical attachment loss | 29-32 weeks of gestation
Bleeding following periodontal probing | 29-32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Panos Papapanou, DDS, PhD, Study Director — Harlem Hospital; Anthony DiAngelis, DMD, Study Director — Hennepin County Medical Center, Minneapolis; William Buchanan, DDS, Study Director — Jackson Medical Mall; John Novak, DDS, Study Director — University of Kentucky
Locations (1):
- Univerisity of Minnesota School Of Dentistry, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Michalowicz BS, Hodges JS, DiAngelis AJ, Lupo VR, Novak MJ, Ferguson JE, Buchanan W, Bofill J, Papapanou PN, Mitchell DA, Matseoane S, Tschida PA; OPT Study. Treatment of periodontal disease and the risk of preterm birth. N Engl J Med. 2006 Nov 2;355(18):1885-94. doi: 10.1056/NEJMoa062249. PMID 17079762